CLINICAL TRIAL: NCT04490044
Title: Under & Over: A Controlled Study to Develop an Upper Limb Rehabilitation Tool for People With Multiple Sclerosis.
Brief Title: Under and Over Rehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Roche Pharma AG (Industry); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 285101
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
Keywords: rehabilitation; design
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Following enrolment and baseline testing participants will be randomised into one of three study arms (Arm 1, Arm 2, Arm 3) and emailed instructions on how to proceed.
Who Masked: Investigator
Masking Description: Randomisation will be done by the researcher and will be blinded to participants' identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): Participants in Arm 1 will be posted the Under & Over study pack (1) and asked to complete the Under & Over tool daily for up to 30 minutes per day, 5 days per week for 3 months. They will be instructed to follow the instruction booklet and complete each pattern in the specific order described in the booklet.
  Interventions: Other: Under & Over rehabilitation tool
- 2 (Active Comparator): Participants in Arm 2 will be posted the Under & Over study pack (2) and asked to complete the Under & Over tool daily for as long or short as they choose or are able to. They will be asked to complete 5 days per week for 3 months. They will be instructed to follow the instruction booklet in any order they wish, choosing which pattern they would like to complete. They will also be encouraged to create their own patterns. These participants will have access to a section of the study website where they will be able to upload photographs of their patterns and see other participants' patterns over the 3-month period.
  Interventions: Other: Under & Over rehabilitation tool
- 3 (Placebo Comparator): Participants in Arm 3 will be posted the Under & Over study pack (3). For the first three months of the study they will be asked to complete the c9HPT 5 days a week. After three months, they will be able to complete the Under & Over tool daily for as long or short as they choose. Similar to Arm 2, They will be asked to do this 5 days per week for 3 months. They will be instructed to follow the instruction booklet in any order they wish, choosing which pattern they would like to
  Interventions: Other: Under & Over rehabilitation tool

INTERVENTIONS:
Other: Under & Over rehabilitation tool — Under & Over is a tool consisting of a 40cm x 40cm white plastic board, two coloured laces and a series of patterns to complete. It enables people to create patterns by threading each lace under, and over the board. It has been designed and developed with people whose upper limb function is affected by their MS. Administration time can be dependent on the person completing it.

SUMMARY:
Multiple Sclerosis (MS) is a progressive neurological condition of the central nervous system for which there is no cure. Symptoms include motor and sensory dysfunction, bladder and bowel dysfunction as well as speech and swallowing difficulties. It commonly leads to cumulative, mixed disabilities over time. The combination of different symptoms and disabilities often limits a person's ability to perform activities of daily living and to actively participate in social and occupational activities which then impacts on their quality of life.

The two main strategies for managing MS symptoms include, medication and rehabilitation. However, historically treatment strategies have focused predominantly on preserving lower limb function thus strategies to improve upper limb function is often neglected. The importance of maintaining upper limb (hand and arm) function is significant for people who have already lost lower limb function. Further loss of functioning contributes to low mood, reduced independence and quality of life.

This study aims to research how an engaging everyday activity, Under & Over, can become a rehabilitation tool to improve upper limb function in people with MS. The study will use a randomised wait list control group design, meaning that participants will be randomised to either the immediate rehabilitation group or the wait list group. Each group will perform the Under & Over task for 12 weeks, following a predetermined programme of instructions. Participants will complete a number of baseline measures measuring their current upper limb function, their quality of life and level of fatigue. This will happen at the start of the study, after 12 weeks of rehabilitation activity and again at a 12 week follow up.

DETAILED DESCRIPTION:
MS is a chronic progressive disease of the central nervous system and is the leading cause of non-traumatic disability in young and middle aged adults. It commonly leads to cumulative, mixed disabilities over time, ranging from motor and sensory impairments to fatigue, impaired vision, cognitive deficits, speech and swallowing problems, bladder, bowel and sexual dysfunction. The combination of different symptoms and disabilities often limits a person's ability to perform activities of daily living and to actively participate in social and occupational activities which then impacts on their quality of life.

Historically, MS treatments have predominantly focused on preserving lower limb function - the ability to walk - and this is reflected in the main areas of clinical practice and research.

Firstly, within the current treatment options, none are licensed for people with advanced forms of MS. Secondly, wheelchair users are excluded from the majority of clinical trials as it is thought to be difficult to measure clinical change in people whose motor functions are already severely affected. Finally, and related to the second point, the gold standard of disease measurement, the expanded disability status scale (EDSS) is weighted towards mobility i.e. a person's ability to walk. Results of a recent study (ASCEND, NCT01416181) highlighted these problems as the primary outcome of the trial was negative; the EDSS and 25-foot timed foot walk, measures of lower limb function dominated the composite measure. However, the nine hole peg test (9HPT), a measure of upper limb function, was positive; trial participants who received natalizumab showed no loss of upper limb function, confirmed at 12 weeks, compared to participants with secondary progressive MS who received placebo.

The Barts MS Research team based at QMUL feel that there now needs to be a shift in focus to reposition the importance of upper limb functions for people with MS.

In August 2016 the investigators launched the #ThinkHand campaign to raise awareness and also initiate discussions amongst patients, clinicians, charities, pharmaceutical companies, regulators and the general public to realise the importance and work towards generating evidence to develop treatments for advanced MS. As part of this campaign, our team has conducted a number of PPI activities at academic conferences, online and at patient events around this topic. Part of this included an online survey where 88% of people with MS (314 of 360 respondents) described their upper limb function to be more important to them than their lower limb function (Dubuisson, Baker, et al., 2017).

This highlights the importance of upper limb function from the patient perspective and the unique experiential knowledge of living with the condition that people with MS have. This is supported by clinical studies; Bertoni et al. (2015) provide evidence that 75% of people with MS have bilateral impaired manual dexterity even in the early stages of the disease. Arm and hand function, are very important to perform activities of daily living like eating, dressing and grooming (Yozbatiran et al., 2006), and even more so for people who have already lost lower limb function as further loss of functioning contributes to low mood, reduced independence and quality of life. Therefore, it is imperative that treatments are aimed at preserving upper limb function.

Tools to maintain upper limb function for people with multiple sclerosis

Current rehabilitation tools and activities focus on measures of body functions and structures looking at the capacity to assess the maximal ability to complete a task or an action (e.g. the 9HPT is gold standard objective measure for manual dexterity (Fischer et al., 1999)) or an activity performance measure measuring the person's habitual performance of tasks in their normal environment (the ABILHAND).

There are a range of upper limb rehabilitation tools in use, but few have been used in MS research and the investigators are aware of only one developed specifically for people with MS (Lamers et al., 2016). For example the ABILHAND was originally developed for rheumatoid arthritis with subsequent versions developed for people with stroke (Penta et al., 1998).

Although these have been validated for use with people with MS (Barrett et al., 2013) their transference from one condition to another poses problems in that the activities that are included lack relevance to the activities specific to living with MS. They also lack relevance to modern living. For example, they are influenced by the ability to walk and there is no mention of urinary catheters, and no mention of new technologies such as the use of touchscreen phones or tablets in the ABILHAND.

Developing a new rehabilitation tool for upper limb function in MS

This study will develop a new upper limb rehabilitation tool to specifically improve upper limb function in people with MS using a more participatory approach to tool development. This is inspired by participatory research as the study has been designed by people with MS and will involve people with MS with upper limb problems, who are the people whose activities are under study.

Outcome measures and rehabilitation activities are typically derived by clinicians and University researchers who only involve patients at specific stages. They therefore embed what these medical and academic professionals believe to be a "good" outcome, i.e. one that is clinically meaningful from the perspective of the clinician and the researcher but these outcomes may not be meaningful to the patients themselves. Further, Lamers and Feys (2014) state that a key characteristic of outcome measures that has been overlooked in MS is how they can be used to facilitate the evolution of rehabilitation content and strategies. This highlights the need to develop tools that include activities that are meaningful to individual patients and can enable them to develop strategies and continue to do these activities.

ELIGIBILITY:
Inclusion Criteria:

* Being able to give online informed consent.
* Over the age of 18. There is no upper age limit.
* Have been diagnosed with Multiple Sclerosis more than 6 months ago and have an Expanded Disability Status Scale (EDSS) of over 6.0 as measured using the online webEDSS
* Understand and be able to communicate (read and write) in English
* Ability to use a computer and access the study resources on the internet

Exclusion Criteria:

* Participants will be ineligible to participate if any inclusion criteria are not met.
* Patients unable to use their hands because of pain or anything that would interfere with the ability to complete the study interventions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Cardboard 9 Hole Peg Test speed at 6 months. | Baseline and 6 months
  The primary outcome measure will be the self-administered Cardboard Nine Hole Peg Test (c9HPT), the raw scores are times to complete the standard task used in the assessment. The aim is to determine if repeated use of the Under & Over tool can improve upper limb function for people with MS using the cardboard nine hole peg test. Raw 9HPT times are skewed rather than normal (Gaussian), but transforming the task times by taking their reciprocal (1/time) leads to an approximately normally distributed measure, and in this form 9HPT is standardly analysed. This reciprocal is readily interpreted as task speed: e.g. if a patient takes 25 seconds to complete the task, the reciprocal, 0.04, is the fraction of the 9HPT task achieved in one second, ie. 4%.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom